CLINICAL TRIAL: NCT06093035
Title: Analysis of Urinary, Vaginal and Intestinal Microbiota in Patients With Neurogenic Bladder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5931
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with neurogenic bladder: Female patients of childbearing age with neurogenic bladder secondary to spina bifida and multiple sclerosis
- healthy patients: Female patients of childbearing age without neurogenic bladder secondary to spina bifida and multiple sclerosis

SUMMARY:
The neurogenic bladder and bowel are two pathological conditions occurring when damaged innervation results in functional alteration of both the bladder and the bowel with a clinical presentation that can vary from retention to incontinence often associated with an increased risk of infection. Specific microbiological patterns of urinary microbiota are associated with states of well-being of the host and play protective and preventive functions for numerous urological pathologies such as urinary tract infections, urinary incontinence and bladder tumors. What the "healthy" profile of the bladder microbiota is in subjects with neurogenic bladder appears currently poorly reported in literature data. Indeed, in these populations different strains of uropathogenic microorganisms, such as E.Coli, Klebsiella, Pseudomonas and Enterococcus, are dominant compared to healthy subjects where Lactobacillus predominates. The characterization of the gut microbiota in terms of composition can be a key tool for understanding the effects that preventive therapeutic and nutritional approaches or clinical procedures have on it, subsequently offering the possibility of improving and complementing these treatments.

Among human microbiota, the vaginal one, the "vaginoma", is among the most studied for its correlation with female health status. The "core" of the vaginal microbiome is Lactobacillus which under physiological conditions is represented in particular by Lactobacillus Crispatus, Lactobacillus Iners, Lactobacillus Jensenii and Lactobacillus Gasseri. Immune cells and related PRRs receptors interact with the microorganisms in the vaginal environment of the vaginal environment are the immune cells and the related PRRs receptors thus the close relationship between microbiome and immunity as well as between vaginoma and genitourinary well-being is now evident. The characterization of the gut, urinary and vaginal microbiota in patients with neurogenic bladder secondary to spina bifida and multiple sclerosis can help identify a "health promoting" profile to personalize and characterize the therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

For both populations:

* childbearing age
* no antibiotic therapies in the last 30 days
* no urinary tract infections/diseases in the last 30 days
* no surgical interventions in the last 90 days
* no intake of prebiotics or probiotics in the last 60 days
* no estrogen-progestin or steroid hormone therapy in the last 60 days
* no sexual intercourse in the last 3 days
* no local vaginal therapy in the last 60 days
* signing of the informed consent;
* patients without lower urinary tract disorders (only for the control group);
* patients with neurogenic bladder secondary to spina bifida (only for the study group).

Exclusion Criteria:

For both populations:

* kidney or urinary tract stones
* presence of pre-existing or ongoing intestinal pathologies (Inflammatory Bowel Diseases, chronic hepatitis, celiac disease, neoplasms, previous extensive intestinal resections)
* ongoing diarrhea of any origin (defined as more than 6 evacuations of watery stools per day and/or faecal volume in 24 hours greater than 250 ml)
* ongoing septic status
* state of pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients of childbearing age with/without neurogenic bladder secondary to spina bifida and multiple sclerosis.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of the urinary vaginal and intestinal microbiome | one day
  Characterization of the urinary vaginal and intestinal microbiome in female patients of reproductive age with neurogenic bladder secondary to spina bifida and multiple sclerosis